CLINICAL TRIAL: NCT04336436
Title: The Impact of Combined Mindfulness-Based Interventions and Nutritional Counseling on Physician Burnout: A Clinical Trial
Brief Title: The Impact of Combined Mindfulness-Based Interventions and Nutritional Counseling on Physician Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1378
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: All participants will receive mindfulness based training and nutritional consultation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Training and Nutrition Counseling (Experimental): Baseline and 3-6 month follow up visits will be arranged for all participants.
  Visits will be conducted at baseline prior to initiation of mindfulness training and nutrition counseling, and at the 3-6 month follow up. Clinical and laboratory assessments will be obtained at each visit.
  Interventions: Behavioral: Mindfulness training; Behavioral: Nutritional consult

INTERVENTIONS:
Behavioral: Mindfulness training — Mindfulness training
Behavioral: Nutritional consult — Nutrition counseling and development of a personalized nutrition plan

SUMMARY:
This study is designed to tackle the issue of physician burnout via a wide-lens approach, integrating both mindfulness-based training and nutritional counseling in the management of professional burnout. The investigators will evaluate the effects of mindfulness training and nutritional counseling interventions through assessment of changes in physiological and biochemical parameters known to be adversely affected in burnout, in addition to the standardized Professional Fulfillment inventory scores at 3-6 months post-intervention.

DETAILED DESCRIPTION:
There is a preponderance of data to support the detrimental effects of burnout on physicians' health and wellbeing. Physician burnout is defined as severe emotional exhaustion, depersonalization towards others and reduced sense of personal achievement. Burnout is often accompanied by feelings of moral distress, loss of interest and energy, and detachment from patients, colleagues and personal relatives. With the recent rapid expansion in global healthcare systems in response to societal changes, rates of physician burnout have been on the rise. It is estimated that 54% of physicians in the United States suffer from professional burnout, a 2-fold higher prevalence than that estimated for the general working population of 28%.

Burnout has serious negative implications on the physical health and wellbeing of individuals. In recent studies, burnout was associated with higher incidence of coronary heart disease and hospitalization from cardiovascular causes. Additionally, burnout was found to be an independent risk factor for type 2 diabetes mellitus and hypercholesterolemia (total cholesterol ≥220 mg/dl). Higher incidence of musculoskeletal pain and pain-related disability were also reported amongst subjects with high burnout. Excessive fatigue, insomnia, headaches, gastrointestinal and respiratory issues were all positively correlated with burnout level. More strikingly, burnout was found to be a significant predictor of mortality in those below the age of 45-years.

Burnout carries its repercussions on mental health as well. In a study of 2,555 dentists, burnout was a significant predictor of depression occurrence during the 3-year follow-up period. Increased psychotropic and antidepressant use was associated with high burnout, with a stronger correlation observed for men than women. High level of burnout was also linked to increased risk of anxiety, substance abuse, alcohol abuse, and even suicidal ideation.

Burnout is a serious threat to the medical profession at large. With more than half of the US physicians suffering from professional burnout, its implications ripple through the entirety of the healthcare system. Burnout decreases both patient care quality and physician productivity. Increased sickness absences have been reported in high burnout. In a recent report, severe burnout independently accounted for 52 sickness absences in a 2-year follow-up period. Additionally, burnout has resulted in more physicians leaving practices or reducing their work hours. A healthcare system loses on average $500,000 to $1,000,000 with the departure of a physician, in addition to the ever-increasing workload of physicians who remain in practice. Most significant of all, burnout leads to major medical errors. With the estimated 250,000 deaths in the United States occurring due to medical errors, developing effective strategies to eliminate physician burnout has become an ever-present priority.

A number of prospective studies and clinical trials have been conducted to assess the efficacy of different interventions on mitigating physician burnout. A major cluster of these studies have focused on behavioral interventions, more specifically, mindfulness-based approaches aimed at reducing the mental and emotional repercussions of burnout. Such behavioral interventions included practices of contemplation-meditation exercises, discussions on enhancing self-care and intensification of present-moment awareness. Efficacy in the latter studies was mostly assessed via quantification of change in burnout and stress-related scores, most notably the Maslach Burnout Inventory score, a well-established tool for assessment of burnout in the occupational setting. The majority of these studies reported favorable effects on burnout scores. However, limited to no-data exist on the physiological and biochemical effects of mindfulness-based interventions on physician burnout.

A second cluster of studies implemented lifestyle changes, more specifically, incentivized exercise programs and nutritional counseling for burnout. However, studies examining the effects of physical activity tended to be short in duration, of small magnitude, and lacked adequate assessment of the physiological and biochemical effects of exercise on burnout [23]. Additionally, a significant lack of research on nutritional and dietary interventions in physician burnout exist in the literature, despite the vitality of good nutrition in the health and wellbeing of physicians.

Therefore, this study intends to tackle the issue of physician burnout via a wide-lens approach, integrating both mindfulness-based training and nutritional counseling in the management of professional burnout. The effects of the interventions will be evaluated through assessment of changes in physiological and biochemical parameters known to be adversely affected in burnout, in addition to the standardized Professional Fulfillment Inventory, at 3-6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physician employed by Cleveland Clinic
* Located in Ohio
* Must anticipate remaining employed for at least 6 months post-enrollment

Exclusion Criteria:

* Non-MD or non-DO healthcare providers
* Unable to commit to intervention sessions
* Current diagnosis of uncontrolled hypertension, and/or uncontrolled diabetes mellitus (defined as hemoglobin A1c ≥9%)
* Current or previous history of Cushing's disease or pheochromocytoma/paraganglioma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Professional Fulfillment Index (PFI) score | 3-6 months
  Measured at baseline and at 3-6 months for each participant to determine if intervention was effective. A higher score indicates improvement.
Change in Neff Self-Compassion Scale score | 3-6 months
  Measured at baseline and at 3-6 months for each participant to determine if intervention was effective. A higher score indicates improvement.

SECONDARY OUTCOMES:
Blood pressure | 3-6 months
  Change in diastolic and systolic blood pressure between baseline and 3-6 months after intervention
Resting heart rate | 3-6 months
  Change in resting heart rate between baseline and 3-6 months after intervention
Weight | 3-6 months
  Change in weight between baseline and 3-6 months after intervention
Athens Insomnia Scale | 3-6 months
  Change in insomnia scale between baseline and 3-6 months after intervention. Range from 0-24 with lower score being favorable outcome.
Daily average time spent reviewing electronic health records | 3-6 months
  Self reported time spent (in hours) reviewing electronic health records
Total Cholesterol | 3-6 months
  Change in total cholesterol post-intervention
Hemoglobin A1c | 3-6 months
  Change in HbA1c post-intervention
Fasting plasma glucose | 3-6 months
  Change in fasting plasma glucose post-intervention
Fasting insulin | 3-6 months
  Change in fasting insulin value post-intervention
C-reactive protein | 3-6 months
  Change in C-reactive protein levels post-intervention
Insulin Resistance | 3-6 months
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) to assess presence of and extent of insulin resistance
High density lipoprotein (HDL) | 3-6 months
  Change in HDL value post-intervention
Low density lipoprotein (LDL) | 3-6 months
  Change in LDL value post-intervention
Triglycerides | 3-6 months
  Change in triglycerides post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Betul Hatipoglu, MD, Principal Investigator — Staff Physician
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahola K, Hakanen J. Job strain, burnout, and depressive symptoms: a prospective study among dentists. J Affect Disord. 2007 Dec;104(1-3):103-10. doi: 10.1016/j.jad.2007.03.004. Epub 2007 Apr 19. PMID 17448543
- [Background] Fred HL, Scheid MS. Physician Burnout: Causes, Consequences, and (?) Cures. Tex Heart Inst J. 2018 Aug 1;45(4):198-202. doi: 10.14503/THIJ-18-6842. eCollection 2018 Aug. No abstract available. PMID 30374225
- [Background] Rothenberger DA. Physician Burnout and Well-Being: A Systematic Review and Framework for Action. Dis Colon Rectum. 2017 Jun;60(6):567-576. doi: 10.1097/DCR.0000000000000844. PMID 28481850
- [Background] Pantenburg B, Luppa M, Konig HH, Riedel-Heller SG. Burnout among young physicians and its association with physicians' wishes to leave: results of a survey in Saxony, Germany. J Occup Med Toxicol. 2016 Jan 22;11:2. doi: 10.1186/s12995-016-0091-z. eCollection 2016. PMID 26807138
- [Background] Dyrbye L, Shanafelt T. A narrative review on burnout experienced by medical students and residents. Med Educ. 2016 Jan;50(1):132-49. doi: 10.1111/medu.12927. PMID 26695473